## Vacuum vs Manual Drainage During Unilateral Thoracentesis Statistical Analysis Description

NCT 03496987

**Original Document Date: 3/2/18** 

Demographic and patient characteristics were compared between participants randomized to the two aspiration methods. Continuous variables were compared using t-tests and categorical variables with chi-square or Fisher's exact statistics. Rates of all-cause complications and early termination of the procedure for each aspiration type were estimated using intercept only negative binomial regression and comparisons of these rates were evaluated using Fisher's exact test. After adjustment for exudative effusion, loculation, malignancy, and recent cardiac procedure, multivariable linear regression evaluated associations between aspiration method and the following four outcomes: change in pain score, total drainage time in seconds, total volume removed in mL, and rate of removal (seconds per 100 mL). All analyses were performed using SAS V9.4 with statistical significance defined as a two-tailed p-value < 0.05.